CLINICAL TRIAL: NCT03758534
Title: The Natural History of Generalized Arterial Calcification of Infancy (GACI) With or Without Autosomal Recessive Hypophosphatemic Rickets Type 2 (ARHR2) or Pseudoxanthoma Elasticum (PXE)
Brief Title: Natural History of GACI With or Without ARHR2 or PXE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität Münster (Other)
Collaborators: ICON plc (Industry)
Responsible Party: Principal Investigator, Frank Rutsch, Prof. Dr. Frank Rutsch, MD, Universität Münster
Other Study IDs: GACI Natural History
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Generalized Arterial Calcification in Infancy; Autosomal Recessive Hypophosphatemic Rickets; Pseudoxanthoma Elasticum
MeSH Terms: conditions — Arterial calcification of infancy; Hypophosphatemic Rickets, Autosomal Recessive, 1; Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is a retrospective chart review study.

SUMMARY:
Generalized arterial calcification of infancy (GACI) is an ultra-rare disorder with an estimated birth prevalence of around 1 in 400,000.1 GACI is generally fatal before birth or within the first six months after birth. The cause of death is frequently myocardial infarction or stroke. GACI is strongly associated with inactivating mutations in ectonucleotide pyrophosphate/ phosphodiesterase 1 (ENPP1). Many patients with GACI, including some without an ENPP1 mutation also present with mutations in adenosine triphosphate binding cassette transporter protein subfamily C member 6 (ABCC6). Autosomal recessive hypophosphatemic rickets type 2 (ARHR2) and pseudoxanthoma elasticum (PXE) are believed to be closely related to GACI. ARHR2 is caused by mutations in the ENPP1 gene and PXE is caused by mutations in the ABCC6 gene, with both being observed among patients with GACI. The natural history of GACI and in particular its long term morbidity and mortality are poorly understood. The primary objective of this study is to characterize overall survival among patients with GACI, over time from birth.

DETAILED DESCRIPTION:
Background:

Generalized arterial calcification of infancy (GACI) is an ultra-rare disorder with an estimated birth prevalence of around 1 in 400,000.1 GACI is characterized by extensive arterial calcifications, arterial stenosis, myointimal proliferation and periarticular calcifications. Individuals with GACI also experience calcification in other body areas, such as joints and organs. GACI is generally fatal before birth or within the first six months after birth. The cause of death is frequently myocardial infarction or stroke. GACI is strongly associated with inactivating mutations in ectonucleotide pyrophosphate/ phosphodiesterase 1 (ENPP1); around three quarters of GACI cases investigated had one or several ENPP1 mutations. Many patients with GACI, including some without an ENPP1 mutation also present with mutations in adenosine triphosphate binding cassette transporter protein subfamily C member 6 (ABCC6). Autosomal recessive hypophosphatemic rickets type 2 (ARHR2) and pseudoxanthoma elasticum (PXE) are believed to be closely related to GACI. ARHR2 is caused by mutations in the ENPP1 gene5 and PXE is caused by mutations in the ABCC6 gene,3 with both being observed among patients with GACI. The natural history of GACI and in particular its long term morbidity and mortality are poorly understood, but a strong understanding of the condition will be crucial for further therapy development and drug testing. This study aims to address this knowledge gap.

Objectives:

The primary objective of this study is to characterize overall survival among patients with GACI, over time from birth.

Secondary objectives are to:

* Characterize the patient and disease characteristics;
* Describe symptomology at diagnosis and the change in symptomology over time;
* Describe treatment patterns specific to GACI or rickets
* Characterize mental/physical impairment, education, and employment situation;
* Characterize the sequelae of the disease;
* Prevalence of rickets; and
* Growth velocities.

Eligibility:

* GACI genotype (mutation in ENPP1 and/or ABCC6) confirmed through mutational analysis of the patient and a GACI phenotype confirmed by imaging or biopsy; or
* GACI phenotype confirmed with imaging, biopsy, or mutational analysis of the parents indicating a GACI genotype (mutation in ENPP1 and/or ABCC6) coinciding with symptoms of the patient.

Data will be collected for both living and deceased patients

Design:

Retrospective multicenter chart review

ELIGIBILITY:
Inclusion Criteria:

* GACI genotype (mutation in ENPP1 and/or ABCC6) confirmed through mutational analysis of the patient and a GACI phenotype confirmed by imaging or biopsy; or
* GACI phenotype confirmed with imaging, biopsy, or mutational analysis of the parents indicating a GACI genotype (mutation in ENPP1 and/or ABCC6) coinciding with symptoms of the patient.
* Data will be collected for both living and deceased patients

Exclusion Criteria:

* Caregivers are not able to give written consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Probands with proven history of generalized arterial calcification of infancy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | Recruitment for this study will end in March 2019
  This study will record the survival rate in patients with GACI

CONTACTS AND LOCATIONS:
Overall Officials: Frank Rutsch, MD, Principal Investigator — WWU Munster
Locations (1):
- WWU Munster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No